CLINICAL TRIAL: NCT01779622
Title: Rapid Versus Slow Ingestion of Mixed Meal: Influence on Islet and Incretin
Brief Title: Rapid Versus Slow Ingestion of Mixed Meal: Influence on Islet and Incretin Hormone Secretion in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Bo Ahren, Professor, Lund University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17; 2013-000449-38 (EudraCT Number)
Record Dates: First submitted 2013-01-27; First posted 2013-01-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Healthy Volunteers Recruited From the General Population
Keywords: mixed meal¨; insulin; glucagon; GIP; GLP-1
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Healthy volunteers are ingesting a mixed meal either rapidly or slowly
  Interventions: Other: Mixed meal

INTERVENTIONS:
Other: Mixed meal — Ingestion of mixed meal

SUMMARY:
To test the influence of rapid versus slow ingestion of a mixed meal on insulin and incretin hormone secretion in healthy volunteers

DETAILED DESCRIPTION:
A mixed meal (524 kcal) is ingested rapidly (within 5 min) or slowly (10-15 min) and changes in insulin, glucagon, GIP and GLP-1 levels are followed for subsequent 300 min

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Diabetes Liver disease Kidney disease Thyroid disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve for insulin | 300 min

SECONDARY OUTCOMES:
Area under the curve for glucose-dependent insuinotropic polypeptide | 300 min
Area under the curve for glucagon-like peptide-1 | 300 min

OTHER OUTCOMES:
Area under the curve for glucagon | 300 min

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Sciences, Lund University, Lund, Sweden

REFERENCES:
- See also: Faculty of Medicine, Lund university — http://www.med.lu.se